CLINICAL TRIAL: NCT00600483
Title: A Randomized, Controlled, Phase 3 Study of Gentamicin-Collagen Sponge in Cardiac Surgical Subjects at Higher Risk for Sternal Wound Infection
Brief Title: Safety and Efficacy of an Antibiotic Implant in Cardiac Surgical Subjects at Higher Risk for Sternal Wound Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Innocoll (Industry)
Collaborators: Duke University (Other); Premier Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: INN-SWI-001
Record Dates: First submitted 2008-01-02; First posted 2008-01-25 (Estimated); Results first posted 2022-05-05 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Cardiac Surgery; Sternal Wound Infection
Keywords: obesity; diabetes
MeSH Terms: conditions — Obesity; Diabetes Mellitus | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- gentamicin Group (Experimental): Insertion of 2 gentamicin-collagen sponges between the sternal halves before closure of the sternotomy
  Interventions: Drug: gentamicin-collagen sponge dipped in saline
- Control Group (No Intervention): Standard of care, ie, insertion of no gentamicin-collagen sponge.

INTERVENTIONS:
Drug: gentamicin-collagen sponge dipped in saline — 100-cm2 sponge
  Arms: gentamicin Group

SUMMARY:
The purpose of this study is to determine whether the gentamicin-collagen sponge is safe and effective in preventing sternal wound infections in patients undergoing cardiac surgery who are at a greater risk of developing sternal wound infections.

DETAILED DESCRIPTION:
Sternal wound infection (SWI) is a significant problem in cardiac surgical subjects,in particular in those with risk factors such as diabetes and obesity. There is a long unmet need for an intervention that can reduce the incidence and severity of SWIs in high-risk subjects.

Gentamicin is an antibiotic that is effective in treating certain kinds of infection. Collagen is a protein that is found in all mammals. The gentamicin-collagen sponge is a thin flat sponge made out of collagen that comes from cow tendons and containing gentamicin. When inserted into a surgical site, the collagen breaks down and the gentamicin is released at the site but very little is absorbed into the blood stream. The high levels of antibiotic at the surgical site may prevent an infection at the surgical site.

Outside of the United States more than 3,500 subjects have received treatment in clinical studies with the gentamicin-collagen sponge, primarily for orthopedic, intraabdominal, and cardiothoracic surgeries or wound infections following surgical procedures or traumatic events.

In this study, all subjects will be given treatment that is normally given to prevent surgical infections. For subjects randomly assigned to the gentamicin-collagen sponge treatment group, 2 sponges will be placed between the sternal halves during surgery. IMMEDIATELY before insertion of the sponge the surgeon should wet the sponge with saline as shown in the training/certification document. This wet sponge SHOULD BE INSERTED INTO THE STERNUM WITHIN APPROXIMATELY 15 SECONDS (AFTER THIS TIME IT MAY BECOME MORE DIFFICULT TO HANDLE). All subjects will be followed for 90 days after surgery to determine whether they develop a sternal wound infection.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo nonemergent CABG and/or valve repair or replacement surgery through a full median sternotomy. This includes the following eligible procedures: isolated CABG surgery, isolated valve surgery, and combined CABG + valve surgery.
* Be at higher risk for SWI, defined as the presence of diabetes mellitus (treated with either oral agent or insulin) and/or obesity, defined as BMI > 30.
* Have the capacity to understand and sign an informed consent form.
* Are male or female and > 18 years of age.
* If female, be postmenopausal (no menstrual period for a minimum of 1 year), be surgically sterilized and have a negative serum or urine pregnancy test on entry in the study, or agree to use adequate birth control during the study and for 3 months after the administration of study agent. Medically acceptable contraceptives include: (1) approved hormonal contraceptives (such as birth control pills, Depo-Provera, or Lupron Depot), (2) barrier methods (such as a condom or diaphragm) used with a spermicide, or (3) an intrauterine device (IUD).
* Agree to be available for evaluation from baseline until final evaluation at 90 days postsurgery.

Exclusion Criteria:

* Known history of hypersensitivity to gentamicin or bovine collagen.
* Undergoing emergency cardiac surgery (urgent surgery is allowed if informed consent is obtained and the study procedures can be performed).
* Undergoing a significant concomitant surgical procedure (eg, carotid endarterectomy, aortic root repair or replacement, DHCA, or pulmonary resection).
* Undergoing a minimally invasive or a thoracic surgical approach.
* Using a preoperative mechanical assist device or IABP if inserted for shock/low output syndrome (an IABP is allowed if it is inserted for unstable angina).
* Active and significant systemic infection, eg active endocarditis, or a history of significant recurrent systemic infection.
* Receiving antibiotic therapy within the 2 weeks before the date of surgery.
* Preoperative serum creatinine > 3 mg/dL or renal failure requiring dialysis.
* History of malignancy within the past year (except for squamous or basal cell carcinoma of the skin that has been treated with no evidence of recurrence).
* History of major organ transplantation, including bone marrow transplantation.
* Recent history of significant drug or alcohol abuse.
* Taking systemic immunosuppressive drugs, including steroids (at a dose > 10 mg oral prednisone daily) or a history of a current immunosuppressive condition (eg, symptomatic HIV infection), defined as a CD4 count < 200.
* Scheduled to receive "stress doses" of glucocorticoids (ie, doses > 2 mg/kg/day of methylprednisolone or equivalent).
* Pregnant, lactating, or of childbearing potential not practicing a birth control method with a high degree of reliability (defined in section 3.1).
* Postsurgical life expectancy ≤ 90 days, in the investigator's or sponsor's opinion.
* Refusal to accept medically indicated blood products.
* Current participation or participation within 30 days before the start of this study in another experimental drug or device study, or is currently participating in a study during which the administration of investigational drugs within 90 days is anticipated.
* Has a moderate or severe pectus deformity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1502 (Actual)
Dates: Start 2007-12; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Prior, Study Director — Innocoll
Locations (42):
- United States (42):
  - Birmingham, Alabama
  - Florence, Alabama
  - Pasadena, California
  - San Francisco, California
  - Brandon, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - Augusta, Georgia
  - Maywood, Illinois
  - Springfield, Illinois
  - Fort Wayne, Indiana
  - West Des Moines, Iowa
  - Olathe, Kansas
  - Wichita, Kansas
  - Baltimore, Maryland
  - Salisbury, Maryland
  - Takoma Park, Maryland
  - Springfield, Massachusetts
  - Bay City, Michigan
  - Lansing, Michigan
  - Saginaw, Michigan
  - St Louis, Missouri
  - Omaha, Nebraska
  - New York, New York
  - Durham, North Carolina
  - Gastonia, North Carolina
  - Greenville, North Carolina
  - Raleigh, North Carolina
  - Winston-Salem, North Carolina
  - Akron, Ohio
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Zanesville, Ohio
  - Portland, Oregon
  - Allentown, Pennsylvania
  - Bethlehem, Pennsylvania
  - Philadelphia, Pennsylvania
  - Dallas, Texas
  - Houston, Texas
  - Tomball, Texas
  - Richmond, Virginia
  - Tacoma, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bennett-Guerrero E, Ferguson TB Jr, Lin M, Garg J, Mark DB, Scavo VA Jr, Kouchoukos N, Richardson JB Jr, Pridgen RL, Corey GR; SWIPE-1 Trial Group. Effect of an implantable gentamicin-collagen sponge on sternal wound infections following cardiac surgery: a randomized trial. JAMA. 2010 Aug 18;304(7):755-62. doi: 10.1001/jama.2010.1152. PMID 20716738

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Gentamicin Group | Control Group
Started | 753 | 749
Completed | 717 | 702
Not Completed | 36 | 47
Not completed — Lost to Follow-up | 26 | 47
Not completed — Randomized but not treated | 10 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gentamicin Group | Control Group | Total
Number analyzed (Participants) | 753 | 749 | 1502
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.3 (9.88) | 64.3 (10.50) | 64.3 (10.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 223 | 219 | 442
  Male | 530 | 530 | 1060
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 5 | 5 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 56 | 59 | 115
  White | 688 | 683 | 1371
  More than one race | 4 | 1 | 5
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Surgical Wound Infections From Surgery Through Post-operative Day 90
Description: Efficacy will be evaluated by a comparison between the 2 study groups of the incidence of surgical wound infections that occur within the period from surgery through postop day 90.
Time Frame: 90 days post cardiac surgery
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Gentamicin Group | Control Group
Number analyzed (Participants) | 753 | 749
Participants | 63 | 65

2. Secondary Outcome: Surgically Treated Surgical Wound Infection Postoperative Day 90
Description: Proportion of patients with surgically treated surgical wound infection adjudicated by an independent blinded committee.
Time Frame: 90 days post cardiac surgery
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Gentamicin Group | Control Group
Number analyzed (Participants) | 753 | 749
Participants | 25 | 37

3. Secondary Outcome: Proportion of Patients With Deep Surgical Wound Infections Based on Centers for Disease Control Criteria Adjudicated by an Independent Blinded Committee.
Time Frame: 90 days post cardiac surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Gentamicin Group | Control Group
Number analyzed (Participants) | 753 | 749
Participants | 14 | 19

4. Secondary Outcome: Proportion of Patients With Superficial Surgical Wound Infections Based on Centers for Disease Control Criteria Adjudicated by an Independent Blinded Committee.
Time Frame: 90 days post cardiac surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Gentamicin Group | Control Group
Number analyzed (Participants) | 753 | 749
Participants | 49 | 46

5. Secondary Outcome: Number of Participants Positive for Each Pathogen Culture
Description: Analysis associated with Microbial Pathogens in Adjudicated 90 Day SWI Subjects ME within Per Protocol Population. Any Microbial Pathogens Detected in SWI (ME)
Time Frame: 90 days post cardiac surgery
Population: PP Population: INN-SWI-001)
Measure: Number; unit: participants
Arm/Group | Gentamicin Group | Control Group
Number analyzed (Participants) | 27 | 32
participants
  Acinetobacter calcoaceticus | 1 | 0
  Coagulase-neg staphylococci | 0 | 2
  Enterobacter cloacae | 2 | 1
  Enterococcus faecalis | 1 | 1
  Escherichia coli | 3 | 3
  Group B species streptococcus | 1 | 0
  Klebsiella pneumoniae | 0 | 2
  Klebsiella spp | 1 | 2
  Methicillin-resistant SA | 2 | 1
  Methicillin-sensitive SA | 6 | 2
  Other Specify 1 | 3 | 3
  Proteus mirabilis | 4 | 5
  Providencia stuartii | 1 | 0
  Pseudomonas aeruginosa | 3 | 3
  Serratia marcescens | 2 | 4
  Staphylococcus aureus | 5 | 6
  Staphylococcus capitis | 1 | 0
  Staphylococcus epidermidis | 2 | 7
  Staphylococcus hominis | 0 | 1
  Staphylococcus lugdunensis | 0 | 1
  Staphylococcus xylosus | 0 | 1
  Streptococcus agalactiae | 1 | 0

6. Secondary Outcome: ASEPSIS Score
Description: ASEPSIS Score through 90 days postoperative - To compare antibiotic regimens for their effectiveness in preventing or treating wound sepsis, well-defined criteria for outcome are needed. A method of assessing wound healing has been devised that defines carefully the characteristics to be considered and how they are to be awarded points. Objective criteria are also included in the assessment. Points are given for the need for Additional treatment, the presence of Serous discharge, Erythema, Purulent exudate, and Separation of the deep tissues, the Isolation of bacteria, and the duration of inpatient Stay (ASEPSIS). The higher the points the worse outcome. Maximum Points would be 60. Minimum points would be 0
Time Frame: 90 days post cardiac surgery
Population: ITT population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Gentamicin Group | Control Group
Number analyzed (Participants) | 753 | 749
score on a scale | 1.9 (6.32) | 2.0 (7.18)

7. Secondary Outcome: Rehospitalization for Sternal Wound Infection
Description: Rehospitalization for Sternal Wound Infection - within 90 days postoperatively.
Time Frame: 90 days post cardiac surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Gentamicin Group | Control Group
Number analyzed (Participants) | 753 | 749
Participants | 23 | 24

ADVERSE EVENTS:
Time Frame: 90 days from Randomization.
Description: 10 Subject were randomized but not treated at the sites by error (mis randomized). Therefore the safety population has 10 less participants receiving Gentamicin and 10 additional in the Control
Groups:
- Control Group: Standard of care, ie, insertion of no gentamicin-collagen sponge. Includes patients randomized to Gentamicin but where not treated in the Gentamicin group
Arm/Group | Gentamicin Group | Control Group
All-Cause Mortality (participants affected / at risk) | 19/743 | 27/759
Serious Adverse Events (participants affected / at risk) | 269/743 | 290/759
Other Adverse Events (participants affected / at risk) | 741/743 | 757/759
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gentamicin Group (N=743) | Control Group (N=759)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
Coagulopathy (Blood and lymphatic system disorders) | 5 (5) | 4 (4)
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 4 (4) | 6 (6)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 2 (2) | 1 (1)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 19 (19) | 23 (23)
Atrial flutter (Cardiac disorders) | 12 (12) | 5 (5)
Atrial tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block (Cardiac disorders) | 2 (2) | 2 (2)
Atrioventricular block complete (Cardiac disorders) | 2 (2) | 4 (4)
Bradycardia (Cardiac disorders) | 10 (10) | 5 (5)
Cardiac arrest (Cardiac disorders) | 6 (6) | 6 (6)
Cardiac failure (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 28 (28) | 29 (29)
Cardiac tamponade (Cardiac disorders) | 3 (3) | 5 (5)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 3 (3)
Coronary artery disease (Cardiac disorders) | 0 (0) | 2 (2)
Dressler's syndrome (Cardiac disorders) | 1 (1) | 2 (2)
Intracardiac thrombus (Cardiac disorders) | 0 (0) | 1 (1)
Ischaemic cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Low cardiac output syndrome (Cardiac disorders) | 0 (0) | 2 (2)
Myocardial infarction (Cardiac disorders) | 1 (1) | 4 (4)
Nodal rhythm (Cardiac disorders) | 2 (2) | 0 (0)
Pericardial effusion (Cardiac disorders) | 5 (5) | 7 (7)
Pericarditis (Cardiac disorders) | 1 (1) | 1 (1)
Sick sinus syndrome (Cardiac disorders) | 5 (5) | 8 (8)
Sinus arrest (Cardiac disorders) | 1 (1) | 1 (1)
Stress cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 1 (1) | 5 (5)
Ventricular tachycardia (Cardiac disorders) | 2 (2) | 3 (3)
Atrial septal defect (Congenital, familial and genetic disorders) | 1 (1) | 1 (1)
Gastrointestinal arteriovenous malformation (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3) | 1 (1)
Diabetic gastroparesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Erosive oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 5 (5)
Gastrointestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 4 (4)
Inguinal hernia, obstructive (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 3 (3)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 4 (4) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 1 (1)
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1)
Volvulus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2)
Asthenia (General disorders) | 2 (2) | 3 (3)
Catheter site haemorrhage (General disorders) | 1 (1) | 0 (0)
Generalised oedema (General disorders) | 1 (1) | 1 (1)
Impaired healing (General disorders) | 1 (1) | 1 (1)
Malaise (General disorders) | 1 (1) | 0 (0)
Mechanical complication of implant (General disorders) | 0 (0) | 1 (1)
Multi-organ failure (General disorders) | 4 (4) | 5 (5)
Non-cardiac chest pain (General disorders) | 9 (9) | 7 (7)
Pyrexia (General disorders) | 2 (2) | 0 (0)
Systemic inflammatory response syndrome (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 3 (3) | 2 (2)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 2 (2)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 3 (3)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 9 (9) | 4 (4)
Cholecystitis infective (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
Diabetic foot infection (Infections and infestations) | 1 (1) | 0 (0)
Enterococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Gangrene (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 1 (1)
Incision site cellulitis (Infections and infestations) | 2 (2) | 0 (0)
Incision site infection (Infections and infestations) | 1 (1) | 1 (1)
Lobar pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Lung infection pseudomonal (Infections and infestations) | 0 (0) | 2 (2)
Mediastinitis (Infections and infestations) | 1 (1) | 2 (2)
Osteomyelitis (Infections and infestations) | 0 (0) | 3 (3)
Pneumonia (Infections and infestations) | 5 (5) | 20 (20)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia escherichia (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia klebsiella (Infections and infestations) | 1 (1) | 1 (1)
Postoperative abscess (Infections and infestations) | 1 (1) | 1 (1)
Postoperative wound infection (Infections and infestations) | 17 (17) | 24 (24)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 5 (5) | 8 (8)
Septic shock (Infections and infestations) | 1 (1) | 1 (1)
Small intestine gangrene (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal abscess (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1) | 1 (1)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal mediastinitis (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Tracheobronchitis (Infections and infestations) | 1 (1) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (2) | 3 (3)
Wound infection (Infections and infestations) | 1 (1) | 2 (2)
Wound infection staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cardiac pacemaker malfunction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cardiac procedure complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Complication of device removal (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Confusion postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Delayed recovery from anaesthesia (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Device breakage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Device leakage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Graft thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Incision site haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Incision site pain (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Operative haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Post procedural bile leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural discharge (Injury, poisoning and procedural complications) | 4 (4) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 9 (9) | 10 (10)
Post procedural myocardial infarction (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Postoperative ileus (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Postoperative renal failure (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 5 (5) | 2 (2)
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural hypotension (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Vascular graft complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular graft occlusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Weaning failure (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 2 (2) | 5 (5)
Anticoagulation drug level below therapeutic (Investigations) | 0 (0) | 1 (1)
Blood glucose fluctuation (Investigations) | 1 (1) | 1 (1)
Blood pressure decreased (Investigations) | 1 (1) | 0 (0)
Clostridium difficile toxin test positive (Investigations) | 1 (1) | 0 (0)
International normalised ratio increased (Investigations) | 1 (1) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
Troponin increased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 4 (4) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Lactic acidosis (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Aphasia (Nervous system disorders) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 1 (1)
Cerebral infarction (Nervous system disorders) | 2 (2) | 3 (3)
Cerebrovascular accident (Nervous system disorders) | 7 (7) | 8 (8)
Cognitive disorder (Nervous system disorders) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0)
Embolic stroke (Nervous system disorders) | 1 (1) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Facial paresis (Nervous system disorders) | 1 (1) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic cerebral infarction (Nervous system disorders) | 0 (0) | 2 (2)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 3 (3) | 2 (2)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 2 (2)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 2 (2)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Unresponsive to stimuli (Nervous system disorders) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Disorientation (Psychiatric disorders) | 0 (0) | 1 (1)
Major depression (Psychiatric disorders) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Azotaemia (Renal and urinary disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephropathy toxic (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 3 (3) | 6 (6)
Renal failure acute (Renal and urinary disorders) | 18 (18) | 23 (23)
Renal failure chronic (Renal and urinary disorders) | 0 (0) | 2 (2)
Renal tubular necrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 2 (2) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 12 (12) | 10 (10)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4)
Laryngeal keratotic plaque (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung hernia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Mediastinal haematoma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Mediastinal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 8 (8)
Mediastinal mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 28 (28) | 25 (25)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 9 (9)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (5)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 9 (9)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 25 (25)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 23 (23) | 21 (21)
Aortic dissection (Vascular disorders) | 0 (0) | 1 (1)
Aortic rupture (Vascular disorders) | 1 (1) | 0 (0)
Aortic stenosis (Vascular disorders) | 1 (1) | 0 (0)
Arterial haemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Arterial thrombosis limb (Vascular disorders) | 1 (1) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 5 (5) | 4 (4)
Femoral artery occlusion (Vascular disorders) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 1 (1)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 8 (8) | 10 (10)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 1 (1)
Labile blood pressure (Vascular disorders) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 1 (1)
Peripheral vascular disorder (Vascular disorders) | 2 (2) | 0 (0)
Phlebitis superficial (Vascular disorders) | 1 (1) | 0 (0)
Shock (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gentamicin Group (N=743) | Control Group (N=759)
Anaemia (Blood and lymphatic system disorders) | 320 | 326
Blood disorder (Blood and lymphatic system disorders) | 0 | 1
Coagulopathy (Blood and lymphatic system disorders) | 4 | 1
Haemoconcentration (Blood and lymphatic system disorders) | 1 | 0
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 40 | 51
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 1 | 3
Hypercoagulation (Blood and lymphatic system disorders) | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 2
Leukocytosis (Blood and lymphatic system disorders) | 164 | 154
Leukopenia (Blood and lymphatic system disorders) | 4 | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 1
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 7 | 1
Neutrophilia (Blood and lymphatic system disorders) | 2 | 1
Splenomegaly (Blood and lymphatic system disorders) | 1 | 0
Thrombocythaemia (Blood and lymphatic system disorders) | 3 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 150 | 161
Acute left ventricular failure (Cardiac disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 2 | 1
Angina pectoris (Cardiac disorders) | 4 | 5
Aortic valve incompetence (Cardiac disorders) | 0 | 1
Aortic valve sclerosis (Cardiac disorders) | 0 | 1
Arrhythmia (Cardiac disorders) | 5 | 11
Arrhythmia supraventricular (Cardiac disorders) | 4 | 1
Atrial fibrillation (Cardiac disorders) | 186 | 192
Atrial flutter (Cardiac disorders) | 12 | 24
Atrial hypertrophy (Cardiac disorders) | 0 | 1
Atrial tachycardia (Cardiac disorders) | 1 | 0
Atrioventricular block (Cardiac disorders) | 4 | 5
Atrioventricular block complete (Cardiac disorders) | 2 | 4
Atrioventricular block first degree (Cardiac disorders) | 7 | 12
Atrioventricular block second degree (Cardiac disorders) | 1 | 1
Bifascicular block (Cardiac disorders) | 1 | 0
Bradyarrhythmia (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 22 | 30
Bundle branch block (Cardiac disorders) | 3 | 3
Bundle branch block left (Cardiac disorders) | 2 | 2
Bundle branch block right (Cardiac disorders) | 3 | 4
Cardiac arrest (Cardiac disorders) | 2 | 1
Cardiac failure (Cardiac disorders) | 0 | 2
Cardiac failure congestive (Cardiac disorders) | 36 | 39
Cardiogenic shock (Cardiac disorders) | 1 | 1
Cardiomegaly (Cardiac disorders) | 80 | 62
Cyanosis (Cardiac disorders) | 1 | 2
Dilatation atrial (Cardiac disorders) | 1 | 0
Dressler's syndrome (Cardiac disorders) | 0 | 1
Extrasystoles (Cardiac disorders) | 5 | 5
Intracardiac thrombus (Cardiac disorders) | 1 | 1
Ischaemic cardiomyopathy (Cardiac disorders) | 1 | 0
Left atrial dilatation (Cardiac disorders) | 0 | 1
Left ventricular dysfunction (Cardiac disorders) | 3 | 1
Left ventricular hypertrophy (Cardiac disorders) | 2 | 0
Mitral valve calcification (Cardiac disorders) | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 2 | 1
Myocardial infarction (Cardiac disorders) | 1 | 2
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Nodal arrhythmia (Cardiac disorders) | 3 | 2
Nodal rhythm (Cardiac disorders) | 9 | 15
Palpitations (Cardiac disorders) | 1 | 1
Pericardial effusion (Cardiac disorders) | 15 | 9
Pericardial rub (Cardiac disorders) | 36 | 32
Pericarditis (Cardiac disorders) | 6 | 7
Pulmonary valve incompetence (Cardiac disorders) | 0 | 1
Right atrial dilatation (Cardiac disorders) | 0 | 1
Sick sinus syndrome (Cardiac disorders) | 1 | 0
Sinus arrest (Cardiac disorders) | 0 | 2
Sinus arrhythmia (Cardiac disorders) | 2 | 1
Sinus bradycardia (Cardiac disorders) | 18 | 15
Sinus tachycardia (Cardiac disorders) | 70 | 60
Supraventricular extrasystoles (Cardiac disorders) | 15 | 12
Supraventricular tachycardia (Cardiac disorders) | 10 | 16
Tachycardia (Cardiac disorders) | 33 | 24
Tachycardia paroxysmal (Cardiac disorders) | 9 | 11
Tricuspid valve incompetence (Cardiac disorders) | 0 | 1
Tricuspid valve prolapse (Cardiac disorders) | 0 | 1
Ventricular arrhythmia (Cardiac disorders) | 3 | 1
Ventricular dysfunction (Cardiac disorders) | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 39 | 30
Ventricular fibrillation (Cardiac disorders) | 0 | 1
Ventricular hypokinesia (Cardiac disorders) | 1 | 1
Ventricular tachycardia (Cardiac disorders) | 28 | 29
Wolff-parkinson-white syndrome (Cardiac disorders) | 0 | 1
Atrial septal defect (Congenital, familial and genetic disorders) | 0 | 1
Deafness (Ear and labyrinth disorders) | 2 | 1
Hypoacusis (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 7 | 3
Vertigo positional (Ear and labyrinth disorders) | 1 | 0
Endocrine disorders (Ear and labyrinth disorders) | 3 | 0
Adrenal mass (Ear and labyrinth disorders) | 1 | 0
Hypothyroidism (Ear and labyrinth disorders) | 2 | 0
Eye disorders (Ear and labyrinth disorders) | 19 | 9
Diplopia (Ear and labyrinth disorders) | 1 | 1
Dry eye (Ear and labyrinth disorders) | 1 | 1
Eye haemorrhage (Ear and labyrinth disorders) | 1 | 1
Eye pruritus (Ear and labyrinth disorders) | 1 | 0
Eye swelling (Ear and labyrinth disorders) | 1 | 1
Lacrimation increased (Ear and labyrinth disorders) | 1 | 1
Myodesopsia (Ear and labyrinth disorders) | 1 | 0
Ocular hyperaemia (Ear and labyrinth disorders) | 1 | 1
Pupils unequal (Ear and labyrinth disorders) | 1 | 1
Retinal artery embolism (Ear and labyrinth disorders) | 1 | 0
Vision blurred (Ear and labyrinth disorders) | 5 | 1
Visual acuity reduced (Ear and labyrinth disorders) | 1 | 1
Visual impairment (Ear and labyrinth disorders) | 2 | 0
Abdominal discomfort (Gastrointestinal disorders) | 9 | 5
Abdominal distension (Gastrointestinal disorders) | 11 | 20
Abdominal pain (Gastrointestinal disorders) | 10 | 5
Abdominal pain lower (Gastrointestinal disorders) | 2 | 2
Abdominal pain upper (Gastrointestinal disorders) | 3 | 2
Abdominal tenderness (Gastrointestinal disorders) | 1 | 1
Ascites (Gastrointestinal disorders) | 1 | 1
Barrett's oesophagus (Gastrointestinal disorders) | 1 | 0
Chapped lips (Gastrointestinal disorders) | 1 | 1
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 134 | 138
Diarrhoea (Gastrointestinal disorders) | 33 | 27
Dry mouth (Gastrointestinal disorders) | 1 | 3
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 10 | 11
Dysphagia (Gastrointestinal disorders) | 8 | 3
Faecal incontinence (Gastrointestinal disorders) | 2 | 4
Faecaloma (Gastrointestinal disorders) | 2 | 0
Flatulence (Gastrointestinal disorders) | 4 | 4
Gastric disorder (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastritis erosive (Gastrointestinal disorders) | 0 | 1
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 1
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 11 | 8
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 1
Gingival bleeding (Gastrointestinal disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 2 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 1
Haemorrhoids (Gastrointestinal disorders) | 2 | 1
Ileus (Gastrointestinal disorders) | 6 | 5
Impaired gastric emptying (Gastrointestinal disorders) | 3 | 2
Intestinal dilatation (Gastrointestinal disorders) | 1 | 0
Lip swelling (Gastrointestinal disorders) | 1 | 1
Melaena (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 254 | 255
Odynophagia (Gastrointestinal disorders) | 1 | 0
Oesophageal ulcer (Gastrointestinal disorders) | 1 | 0
Oral disorder (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 2 | 1
Peptic ulcer (Gastrointestinal disorders) | 1 | 0
Peritoneal haematoma (Gastrointestinal disorders) | 0 | 1
Proctalgia (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 3
Reflux oesophagitis (Gastrointestinal disorders) | 0 | 1
Retching (Gastrointestinal disorders) | 0 | 1
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 | 1
Salivary gland cyst (Gastrointestinal disorders) | 1 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 3 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Stomatitis (Gastrointestinal disorders) | 2 | 0
Swollen tongue (Gastrointestinal disorders) | 1 | 2
Tongue oedema (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 1
Umbilical hernia, obstructive (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 52 | 55
Adverse drug reaction (General disorders) | 1 | 1
Asthenia (General disorders) | 49 | 43
Axillary pain (General disorders) | 1 | 1
Breakthrough pain (General disorders) | 0 | 2
Catheter site discharge (General disorders) | 1 | 2
Catheter site haematoma (General disorders) | 2 | 3
Catheter site haemorrhage (General disorders) | 3 | 5
Catheter site pain (General disorders) | 3 | 2
Catheter site related reaction (General disorders) | 0 | 1
Catheter thrombosis (General disorders) | 0 | 1
Chest discomfort (General disorders) | 3 | 2
Chest pain (General disorders) | 6 | 2
Chills (General disorders) | 11 | 8
Discomfort (General disorders) | 4 | 0
Face oedema (General disorders) | 0 | 1
Fatigue (General disorders) | 15 | 10
Feeling cold (General disorders) | 1 | 0
Feeling hot (General disorders) | 1 | 2
Gait disturbance (General disorders) | 4 | 3
General symptom (General disorders) | 0 | 1
Generalised oedema (General disorders) | 208 | 224
Granuloma (General disorders) | 1 | 0
Hyperthermia (General disorders) | 2 | 0
Hypothermia (General disorders) | 1 | 0
Impaired healing (General disorders) | 3 | 3
Implant site pain (General disorders) | 1 | 0
Inflammation (General disorders) | 0 | 2
Infusion site erythema (General disorders) | 1 | 1
Infusion site extravasation (General disorders) | 3 | 2
Infusion site haemorrhage (General disorders) | 1 | 0
Infusion site inflammation (General disorders) | 0 | 1
Infusion site pain (General disorders) | 4 | 3
Infusion site swelling (General disorders) | 1 | 1
Infusion site ulcer (General disorders) | 0 | 1
Infusion site warmth (General disorders) | 0 | 1
Irritability (General disorders) | 3 | 0
Local swelling (General disorders) | 1 | 2
Localised oedema (General disorders) | 2 | 0
Malaise (General disorders) | 2 | 1
Non-cardiac chest pain (General disorders) | 8 | 14
Oedema peripheral (General disorders) | 136 | 141
Pain (General disorders) | 14 | 24
Pitting oedema (General disorders) | 0 | 1
Pyrexia (General disorders) | 123 | 115
Submandibular mass (General disorders) | 1 | 0
Wound necrosis (General disorders) | 1 | 0
Biliary dyskinesia (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 3 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 2
Hepatic failure (Hepatobiliary disorders) | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1
Hepatic ischaemia (Hepatobiliary disorders) | 0 | 1
Hepatic steatosis (Hepatobiliary disorders) | 0 | 1
Hepatitis acute (Hepatobiliary disorders) | 0 | 1
Hepatomegaly (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Ischaemic hepatitis (Hepatobiliary disorders) | 2 | 2
Jaundice (Hepatobiliary disorders) | 2 | 1
Portal hypertension (Hepatobiliary disorders) | 1 | 0
Immune system disorders (Hepatobiliary disorders) | 5 | 4
Allergic oedema (Hepatobiliary disorders) | 0 | 1
Allergy to chemicals (Hepatobiliary disorders) | 0 | 1
Drug hypersensitivity (Hepatobiliary disorders) | 2 | 0
Hypersensitivity (Hepatobiliary disorders) | 1 | 1
Seasonal allergy (Hepatobiliary disorders) | 2 | 1
Abdominal abscess (Infections and infestations) | 0 | 1
Abscess limb (Infections and infestations) | 1 | 0
Acarodermatitis (Infections and infestations) | 1 | 0
Acute sinusitis (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 1 | 1
Bacterial disease carrier (Infections and infestations) | 0 | 1
Bacteriuria (Infections and infestations) | 1 | 0
Balanitis candida (Infections and infestations) | 0 | 1
Breast abscess (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 14 | 14
Candidiasis (Infections and infestations) | 6 | 2
Candiduria (Infections and infestations) | 0 | 1
Catheter site infection (Infections and infestations) | 1 | 1
Cellulitis (Infections and infestations) | 15 | 16
Clostridial infection (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 3
Cystitis (Infections and infestations) | 1 | 2
Cystitis klebsiella (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 1 | 2
Escherichia bacteraemia (Infections and infestations) | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 2 | 2
Fungal infection (Infections and infestations) | 1 | 0
Fungal skin infection (Infections and infestations) | 2 | 1
Gastroenteritis (Infections and infestations) | 1 | 1
Haemophilus infection (Infections and infestations) | 0 | 1
Helicobacter infection (Infections and infestations) | 1 | 0
Hepatitis b (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 1
Incision site cellulitis (Infections and infestations) | 4 | 3
Incision site infection (Infections and infestations) | 4 | 1
Infection (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 4 | 1
Infusion site infection (Infections and infestations) | 0 | 1
Kidney infection (Infections and infestations) | 0 | 1
Liver abscess (Infections and infestations) | 0 | 1
Lobar pneumonia (Infections and infestations) | 1 | 3
Localised infection (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 1
Lung infection (Infections and infestations) | 0 | 2
Lung infection pseudomonal (Infections and infestations) | 1 | 1
Mastoiditis (Infections and infestations) | 0 | 1
Nail infection (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 2 | 4
Oral candidiasis (Infections and infestations) | 1 | 2
Oral fungal infection (Infections and infestations) | 1 | 0
Oral herpes (Infections and infestations) | 1 | 1
Pharyngitis (Infections and infestations) | 0 | 1
Pharyngitis streptococcal (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 24 | 16
Pneumonia bacterial (Infections and infestations) | 1 | 0
Pneumonia staphylococcal (Infections and infestations) | 1 | 0
Pneumonia streptococcal (Infections and infestations) | 1 | 0
Post procedural cellulitis (Infections and infestations) | 4 | 5
Postoperative wound infection (Infections and infestations) | 12 | 22
Pseudomonas bronchitis (Infections and infestations) | 1 | 0
Purulent discharge (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 3
Rhinitis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 3
Sinusitis (Infections and infestations) | 8 | 8
Skin candida (Infections and infestations) | 2 | 2
Skin infection (Infections and infestations) | 0 | 1
Sputum purulent (Infections and infestations) | 1 | 2
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1
Staphylococcal mediastinitis (Infections and infestations) | 0 | 1
Stitch abscess (Infections and infestations) | 0 | 2
Subcutaneous abscess (Infections and infestations) | 1 | 0
Tinea cruris (Infections and infestations) | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 2
Tracheobronchitis (Infections and infestations) | 2 | 1
Upper respiratory tract infection (Infections and infestations) | 7 | 4
Urinary tract infection (Infections and infestations) | 33 | 48
Urinary tract infection bacterial (Infections and infestations) | 2 | 1
Urinary tract infection pseudomonal (Infections and infestations) | 2 | 1
Vulvovaginal candidiasis (Infections and infestations) | 1 | 1
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 1
Wound infection (Infections and infestations) | 8 | 4
Wound infection pseudomonas (Infections and infestations) | 0 | 1
Agitation postoperative (Injury, poisoning and procedural complications) | 0 | 5
Anaemia postoperative (Injury, poisoning and procedural complications) | 43 | 49
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 1 | 0
Brachial plexus injury (Injury, poisoning and procedural complications) | 0 | 1
Cartilage injury (Injury, poisoning and procedural complications) | 1 | 0
Collapse of lung (Injury, poisoning and procedural complications) | 1 | 0
Confusion postoperative (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 7 | 5
Device breakage (Injury, poisoning and procedural complications) | 1 | 1
Device dislocation (Injury, poisoning and procedural complications) | 1 | 0
Device leakage (Injury, poisoning and procedural complications) | 2 | 2
Endotracheal intubation complication (Injury, poisoning and procedural complications) | 0 | 1
Excoriation (Injury, poisoning and procedural complications) | 6 | 7
Fall (Injury, poisoning and procedural complications) | 1 | 2
Incision site blister (Injury, poisoning and procedural complications) | 1 | 3
Incision site complication (Injury, poisoning and procedural complications) | 0 | 2
Incision site erythema (Injury, poisoning and procedural complications) | 6 | 5
Incision site haematoma (Injury, poisoning and procedural complications) | 1 | 5
Incision site haemorrhage (Injury, poisoning and procedural complications) | 12 | 15
Incision site oedema (Injury, poisoning and procedural complications) | 0 | 2
Incision site pain (Injury, poisoning and procedural complications) | 405 | 419
Incision site pruritus (Injury, poisoning and procedural complications) | 1 | 1
Medical device pain (Injury, poisoning and procedural complications) | 1 | 2
Mental status changes postoperative (Injury, poisoning and procedural complications) | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1
Open wound (Injury, poisoning and procedural complications) | 1 | 0
Operative haemorrhage (Injury, poisoning and procedural complications) | 1 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 3 | 1
Post procedural discharge (Injury, poisoning and procedural complications) | 55 | 58
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 1
Post procedural haematuria (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 8 | 19
Post procedural myocardial infarction (Injury, poisoning and procedural complications) | 2 | 3
Post procedural oedema (Injury, poisoning and procedural complications) | 1 | 0
Postoperative ileus (Injury, poisoning and procedural complications) | 2 | 2
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 4 | 6
Postoperative wound complication (Injury, poisoning and procedural complications) | 11 | 20
Postpericardiotomy syndrome (Injury, poisoning and procedural complications) | 1 | 2
Procedural complication (Injury, poisoning and procedural complications) | 1 | 0
Procedural hypertension (Injury, poisoning and procedural complications) | 1 | 3
Procedural hypotension (Injury, poisoning and procedural complications) | 6 | 7
Procedural nausea (Injury, poisoning and procedural complications) | 1 | 5
Procedural pain (Injury, poisoning and procedural complications) | 182 | 169
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Seroma (Injury, poisoning and procedural complications) | 1 | 3
Skin laceration (Injury, poisoning and procedural complications) | 9 | 8
Surgical skin tear (Injury, poisoning and procedural complications) | 0 | 1
Suture rupture (Injury, poisoning and procedural complications) | 0 | 1
Synovial rupture (Injury, poisoning and procedural complications) | 1 | 0
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0
Thrombosis in device (Injury, poisoning and procedural complications) | 1 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 1 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 1
Urethral injury (Injury, poisoning and procedural complications) | 1 | 0
Urinary retention postoperative (Injury, poisoning and procedural complications) | 0 | 1
Vascular graft occlusion (Injury, poisoning and procedural complications) | 0 | 1
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 | 0
Vasoplegia syndrome (Injury, poisoning and procedural complications) | 1 | 0
Wound (Injury, poisoning and procedural complications) | 3 | 1
Wound complication (Injury, poisoning and procedural complications) | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 9 | 11
Acid base balance abnormal (Investigations) | 1 | 1
Activated partial thromboplastin time prolonged (Investigations) | 2 | 4
Alanine aminotransferase decreased (Investigations) | 2 | 0
Alanine aminotransferase increased (Investigations) | 2 | 1
Ammonia increased (Investigations) | 1 | 0
Anticoagulation drug level below therapeutic (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 9 | 5
Aspiration bronchial (Investigations) | 0 | 1
Bacteria sputum identified (Investigations) | 17 | 8
Bacterial culture positive (Investigations) | 3 | 13
Base excess increased (Investigations) | 1 | 0
Basophil count increased (Investigations) | 0 | 1
Blood albumin decreased (Investigations) | 12 | 9
Blood alkaline phosphatase decreased (Investigations) | 4 | 3
Blood alkaline phosphatase increased (Investigations) | 1 | 0
Blood bicarbonate decreased (Investigations) | 0 | 2
Blood bicarbonate increased (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 3 | 0
Blood calcium decreased (Investigations) | 21 | 19
Blood calcium increased (Investigations) | 1 | 2
Blood chloride decreased (Investigations) | 0 | 2
Blood chloride increased (Investigations) | 7 | 5
Blood cortisol decreased (Investigations) | 0 | 1
Blood creatine increased (Investigations) | 3 | 2
Blood creatine phosphokinase increased (Investigations) | 2 | 2
Blood creatine phosphokinase mb increased (Investigations) | 2 | 0
Blood creatinine decreased (Investigations) | 1 | 1
Blood creatinine increased (Investigations) | 44 | 38
Blood fibrinogen decreased (Investigations) | 1 | 0
Blood glucose fluctuation (Investigations) | 11 | 14
Blood glucose increased (Investigations) | 23 | 26
Blood lactic acid increased (Investigations) | 0 | 5
Blood magnesium decreased (Investigations) | 13 | 6
Blood magnesium increased (Investigations) | 10 | 10
Blood ph decreased (Investigations) | 0 | 2
Blood phosphorus decreased (Investigations) | 2 | 2
Blood phosphorus increased (Investigations) | 2 | 2
Blood potassium decreased (Investigations) | 5 | 4
Blood potassium increased (Investigations) | 5 | 11
Blood pressure decreased (Investigations) | 3 | 5
Blood pressure increased (Investigations) | 5 | 10
Blood pressure systolic decreased (Investigations) | 1 | 0
Blood pressure systolic increased (Investigations) | 1 | 0
Blood sodium decreased (Investigations) | 7 | 8
Blood sodium increased (Investigations) | 2 | 2
Blood thyroid stimulating hormone increased (Investigations) | 2 | 0
Blood urea increased (Investigations) | 38 | 35
Blood urea nitrogen/creatinine ratio increased (Investigations) | 1 | 0
Blood urine present (Investigations) | 1 | 2
Body temperature decreased (Investigations) | 1 | 0
Body temperature increased (Investigations) | 55 | 53
Brain natriuretic peptide increased (Investigations) | 4 | 4
Breath sounds abnormal (Investigations) | 56 | 56
C-reactive protein increased (Investigations) | 1 | 0
Calcium ionised decreased (Investigations) | 21 | 24
Carbon dioxide decreased (Investigations) | 2 | 0
Carbon dioxide increased (Investigations) | 4 | 5
Cardiac enzymes increased (Investigations) | 2 | 3
Cardiac index decreased (Investigations) | 18 | 18
Cardiac murmur (Investigations) | 1 | 1
Cardiac output decreased (Investigations) | 6 | 7
Cardioactive drug level decreased (Investigations) | 1 | 0
Central venous pressure decreased (Investigations) | 5 | 2
Chest x-ray abnormal (Investigations) | 7 | 5
Clostridium difficile toxin test positive (Investigations) | 0 | 1
Computerised tomogram abdomen abnormal (Investigations) | 0 | 1
Ejection fraction decreased (Investigations) | 0 | 2
Electrocardiogram abnormal (Investigations) | 0 | 1
Electrocardiogram st segment depression (Investigations) | 0 | 1
Electrocardiogram st segment elevation (Investigations) | 7 | 8
Fibrin d dimer increased (Investigations) | 0 | 1
Fungus sputum test positive (Investigations) | 0 | 3
Glycosylated haemoglobin increased (Investigations) | 0 | 1
Grip strength decreased (Investigations) | 1 | 0
Haematocrit decreased (Investigations) | 28 | 38
Haemoglobin decreased (Investigations) | 20 | 26
Heart rate decreased (Investigations) | 3 | 2
Heart rate increased (Investigations) | 3 | 2
Heart rate irregular (Investigations) | 1 | 2
Heart sounds abnormal (Investigations) | 1 | 1
Hepatic enzyme increased (Investigations) | 3 | 2
International normalised ratio decreased (Investigations) | 0 | 1
International normalised ratio increased (Investigations) | 3 | 2
Lipase increased (Investigations) | 1 | 0
Liver function test abnormal (Investigations) | 8 | 6
Lymphocyte count decreased (Investigations) | 12 | 7
Mean arterial pressure decreased (Investigations) | 1 | 1
Methicillin-resistant staphylococcal aureus test positive (Investigations) | 2 | 7
Monocyte count increased (Investigations) | 3 | 1
Myoglobin blood increased (Investigations) | 0 | 1
Neutrophil count increased (Investigations) | 8 | 7
Occult blood (Investigations) | 0 | 1
Occult blood positive (Investigations) | 1 | 1
Oxygen saturation decreased (Investigations) | 12 | 8
Platelet count decreased (Investigations) | 13 | 13
Platelet count increased (Investigations) | 3 | 6
Protein total decreased (Investigations) | 8 | 6
Prothrombin time prolonged (Investigations) | 5 | 3
Prothrombin time ratio increased (Investigations) | 0 | 1
Pulmonary arterial pressure decreased (Investigations) | 1 | 1
Pulmonary arterial pressure increased (Investigations) | 2 | 0
Pulmonary arterial wedge pressure increased (Investigations) | 0 | 1
Pulse absent (Investigations) | 0 | 2
Pulse pressure decreased (Investigations) | 0 | 1
Red blood cell count decreased (Investigations) | 11 | 10
Serum ferritin increased (Investigations) | 1 | 0
Sputum abnormal (Investigations) | 0 | 2
Staphylococcal identification test positive (Investigations) | 0 | 2
Streptococcal identification test positive (Investigations) | 1 | 2
Total lung capacity decreased (Investigations) | 2 | 0
Transaminases increased (Investigations) | 1 | 0
Troponin i increased (Investigations) | 0 | 2
Troponin increased (Investigations) | 10 | 5
Urinary sediment present (Investigations) | 1 | 0
Urine analysis abnormal (Investigations) | 0 | 1
Urine colour abnormal (Investigations) | 2 | 0
Urine output decreased (Investigations) | 51 | 65
Vascular resistance systemic decreased (Investigations) | 0 | 1
Vascular resistance systemic increased (Investigations) | 1 | 1
Venous oxygen saturation decreased (Investigations) | 0 | 2
Venous pressure increased (Investigations) | 1 | 0
Weight decreased (Investigations) | 1 | 1
Weight increased (Investigations) | 2 | 0
White blood cell count decreased (Investigations) | 0 | 2
White blood cell count increased (Investigations) | 112 | 105
Acidosis (Metabolism and nutrition disorders) | 3 | 2
Anorexia (Metabolism and nutrition disorders) | 5 | 6
Decreased appetite (Metabolism and nutrition disorders) | 28 | 22
Dehydration (Metabolism and nutrition disorders) | 3 | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 17 | 14
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 3
Fluid overload (Metabolism and nutrition disorders) | 57 | 59
Fluid retention (Metabolism and nutrition disorders) | 3 | 3
Glucose tolerance impaired (Metabolism and nutrition disorders) | 3 | 3
Gout (Metabolism and nutrition disorders) | 1 | 6
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 2
Hyperchloraemia (Metabolism and nutrition disorders) | 3 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 152 | 142
Hyperkalaemia (Metabolism and nutrition disorders) | 73 | 59
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 1
Hypermagnesaemia (Metabolism and nutrition disorders) | 10 | 15
Hypernatraemia (Metabolism and nutrition disorders) | 4 | 9
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 1 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 102 | 98
Hypochloraemia (Metabolism and nutrition disorders) | 3 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 58 | 50
Hypokalaemia (Metabolism and nutrition disorders) | 112 | 130
Hypomagnesaemia (Metabolism and nutrition disorders) | 18 | 19
Hyponatraemia (Metabolism and nutrition disorders) | 47 | 47
Hypophosphataemia (Metabolism and nutrition disorders) | 5 | 6
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 5 | 4
Iron deficiency (Metabolism and nutrition disorders) | 0 | 1
Lactic acidosis (Metabolism and nutrition disorders) | 2 | 1
Malnutrition (Metabolism and nutrition disorders) | 10 | 8
Metabolic acidosis (Metabolism and nutrition disorders) | 11 | 8
Metabolic alkalosis (Metabolism and nutrition disorders) | 1 | 1
Metabolic syndrome (Metabolism and nutrition disorders) | 1 | 2
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 3
Vitamin d deficiency (Metabolism and nutrition disorders) | 3 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 10
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 47 | 35
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Coccydynia (Musculoskeletal and connective tissue disorders) | 1 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 3 | 4
Joint crepitation (Musculoskeletal and connective tissue disorders) | 2 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 | 1
Lower extremity mass (Musculoskeletal and connective tissue disorders) | 2 | 0
Mobility decreased (Musculoskeletal and connective tissue disorders) | 3 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 7
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 14 | 14
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 28 | 27
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 3 | 1
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 27 | 33
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 6
Neck pain (Musculoskeletal and connective tissue disorders) | 9 | 5
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 24 | 33
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 1
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 2
Soft tissue disorder (Musculoskeletal and connective tissue disorders) | 2 | 3
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Aphasia (Nervous system disorders) | 2 | 1
Balance disorder (Nervous system disorders) | 3 | 1
Burning sensation (Nervous system disorders) | 2 | 1
Carotid arteriosclerosis (Nervous system disorders) | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 2 | 0
Cerebellar infarction (Nervous system disorders) | 0 | 1
Cerebral cyst (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 1 | 3
Depressed level of consciousness (Nervous system disorders) | 1 | 2
Dizziness (Nervous system disorders) | 24 | 38
Dizziness exertional (Nervous system disorders) | 2 | 0
Dysarthria (Nervous system disorders) | 1 | 1
Dysgeusia (Nervous system disorders) | 1 | 1
Dysphasia (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 5 | 5
Facial palsy (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 38 | 22
Hemiparesis (Nervous system disorders) | 2 | 2
Hepatic encephalopathy (Nervous system disorders) | 0 | 1
Hyperaesthesia (Nervous system disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 19 | 20
Hypotonia (Nervous system disorders) | 0 | 1
Lethargy (Nervous system disorders) | 16 | 16
Loss of consciousness (Nervous system disorders) | 1 | 0
Memory impairment (Nervous system disorders) | 2 | 1
Metabolic encephalopathy (Nervous system disorders) | 1 | 2
Migraine (Nervous system disorders) | 1 | 0
Nerve compression (Nervous system disorders) | 0 | 1
Neuralgia (Nervous system disorders) | 4 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 3
Paraesthesia (Nervous system disorders) | 4 | 3
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 2 | 1
Restless legs syndrome (Nervous system disorders) | 0 | 1
Sedation (Nervous system disorders) | 0 | 3
Somnolence (Nervous system disorders) | 4 | 2
Syncope (Nervous system disorders) | 2 | 5
Thalamic infarction (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 2
Tremor (Nervous system disorders) | 2 | 3
Unresponsive to stimuli (Nervous system disorders) | 1 | 0
Upper motor neurone lesion (Nervous system disorders) | 1 | 0
Abnormal dreams (Psychiatric disorders) | 0 | 1
Aggression (Psychiatric disorders) | 1 | 1
Agitation (Psychiatric disorders) | 27 | 24
Anxiety (Psychiatric disorders) | 60 | 40
Claustrophobia (Psychiatric disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 57 | 61
Delirium (Psychiatric disorders) | 4 | 3
Depressed mood (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 12 | 11
Disorientation (Psychiatric disorders) | 8 | 5
Hallucination (Psychiatric disorders) | 7 | 6
Hallucination, visual (Psychiatric disorders) | 3 | 7
Insomnia (Psychiatric disorders) | 4 | 52
Mania (Psychiatric disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 12 | 11
Mood altered (Psychiatric disorders) | 1 | 0
Nervousness (Psychiatric disorders) | 0 | 1
Paranoia (Psychiatric disorders) | 1 | 2
Psychotic disorder (Psychiatric disorders) | 1 | 1
Restlessness (Psychiatric disorders) | 16 | 17
Sleep disorder (Psychiatric disorders) | 2 | 1
Stress (Psychiatric disorders) | 0 | 1
Acute prerenal failure (Renal and urinary disorders) | 2 | 0
Anuria (Renal and urinary disorders) | 0 | 1
Azotaemia (Renal and urinary disorders) | 2 | 0
Bladder fibrosis (Renal and urinary disorders) | 1 | 0
Bladder spasm (Renal and urinary disorders) | 2 | 1
Chromaturia (Renal and urinary disorders) | 3 | 5
Dysuria (Renal and urinary disorders) | 11 | 4
Haematuria (Renal and urinary disorders) | 15 | 12
Micturition urgency (Renal and urinary disorders) | 1 | 3
Nephrolithiasis (Renal and urinary disorders) | 3 | 1
Neurogenic bladder (Renal and urinary disorders) | 1 | 0
Nocturia (Renal and urinary disorders) | 1 | 1
Oliguria (Renal and urinary disorders) | 12 | 11
Pollakiuria (Renal and urinary disorders) | 2 | 1
Polyuria (Renal and urinary disorders) | 2 | 1
Proteinuria (Renal and urinary disorders) | 2 | 0
Renal cyst (Renal and urinary disorders) | 1 | 0
Renal disorder (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 60 | 48
Renal failure acute (Renal and urinary disorders) | 26 | 34
Renal failure chronic (Renal and urinary disorders) | 5 | 2
Renal impairment (Renal and urinary disorders) | 1 | 2
Renal mass (Renal and urinary disorders) | 0 | 1
Renal tubular necrosis (Renal and urinary disorders) | 1 | 2
Urinary incontinence (Renal and urinary disorders) | 8 | 13
Urinary retention (Renal and urinary disorders) | 15 | 15
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1
Urine abnormality (Renal and urinary disorders) | 2 | 2
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0
Breast pain (Reproductive system and breast disorders) | 1 | 0
Genital erythema (Reproductive system and breast disorders) | 1 | 0
Genital rash (Reproductive system and breast disorders) | 1 | 0
Penile oedema (Reproductive system and breast disorders) | 0 | 1
Perineal pain (Reproductive system and breast disorders) | 0 | 1
Prostatomegaly (Reproductive system and breast disorders) | 1 | 0
Scrotal erythema (Reproductive system and breast disorders) | 0 | 1
Scrotal haematocoele (Reproductive system and breast disorders) | 1 | 0
Scrotal oedema (Reproductive system and breast disorders) | 1 | 2
Scrotal swelling (Reproductive system and breast disorders) | 1 | 1
Testicular pain (Reproductive system and breast disorders) | 1 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 1 | 0
Vaginal discharge (Reproductive system and breast disorders) | 2 | 1
Acquired diaphragmatic eventration (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 6 | 7
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 270 | 283
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchial oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bullous lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 8 | 3
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 63 | 58
Cough decreased (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Diaphragmatic paralysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 9 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 65 | 60
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 14 | 10
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 8
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 6 | 3
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 48 | 42
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Lung hyperinflation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 18 | 14
Mediastinal disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Mediastinal haematoma (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Mediastinal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal blistering (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 9 | 12
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngeal haematoma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 281 | 277
Pleural rub (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 55 | 46
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 56 | 41
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 65 | 53
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 67 | 73
Pulmonary vascular disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 32 | 19
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 10 | 7
Respiratory alkalosis (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 45 | 32
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 14 | 18
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 7
Wheezing (Respiratory, thoracic and mediastinal disorders) | 27 | 15
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1
Blister (Skin and subcutaneous tissue disorders) | 6 | 10
Cold sweat (Skin and subcutaneous tissue disorders) | 2 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 9 | 8
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 9 | 6
Diabetic bullosis (Skin and subcutaneous tissue disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 10 | 16
Erythema (Skin and subcutaneous tissue disorders) | 9 | 12
Heat rash (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 15 | 10
Hypoaesthesia facial (Skin and subcutaneous tissue disorders) | 1 | 0
Livedo reticularis (Skin and subcutaneous tissue disorders) | 1 | 1
Penile ulceration (Skin and subcutaneous tissue disorders) | 1 | 0
Periorbital oedema (Skin and subcutaneous tissue disorders) | 1 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 9 | 7
Pruritus allergic (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 13 | 15
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1
Skin burning sensation (Skin and subcutaneous tissue disorders) | 1 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 4 | 8
Skin ulcer (Skin and subcutaneous tissue disorders) | 4 | 4
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 5 | 4
Urticaria (Skin and subcutaneous tissue disorders) | 3 | 0
Vascular disorders (Vascular disorders) | 253 | 265
Aortic aneurysm (Vascular disorders) | 0 | 1
Aortic arteriosclerosis (Vascular disorders) | 1 | 0
Blood pressure fluctuation (Vascular disorders) | 2 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 6
Femoral artery aneurysm (Vascular disorders) | 0 | 1
Flushing (Vascular disorders) | 3 | 1
Haematoma (Vascular disorders) | 5 | 5
Haemodynamic instability (Vascular disorders) | 2 | 0
Hypertension (Vascular disorders) | 61 | 68
Hypotension (Vascular disorders) | 182 | 185
Hypovolaemic shock (Vascular disorders) | 1 | 0
Jugular vein thrombosis (Vascular disorders) | 1 | 2
Labile blood pressure (Vascular disorders) | 21 | 14
Labile hypertension (Vascular disorders) | 0 | 1
Lymphocele (Vascular disorders) | 1 | 1
Orthostatic hypotension (Vascular disorders) | 3 | 0
Pallor (Vascular disorders) | 2 | 8
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 2
Peripheral coldness (Vascular disorders) | 2 | 2
Peripheral embolism (Vascular disorders) | 0 | 1
Peripheral ischaemia (Vascular disorders) | 1 | 2
Peripheral vascular disorder (Vascular disorders) | 1 | 0
Phlebitis (Vascular disorders) | 3 | 5
Shock haemorrhagic (Vascular disorders) | 0 | 1
Subclavian artery stenosis (Vascular disorders) | 1 | 0
Subclavian vein thrombosis (Vascular disorders) | 0 | 1
Thrombophlebitis superficial (Vascular disorders) | 3 | 2
Thrombosis (Vascular disorders) | 1 | 1
Vasospasm (Vascular disorders) | 0 | 1
Venous insufficiency (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No